CLINICAL TRIAL: NCT01040936
Title: Intensive Lipid Lowering Treatment in Patients With Non-ST-elevation ACS Undergoing Percutaneous Coronary Intervention
Brief Title: Intensive Lipid Lowering Treatment in Non-ST-elevation Acute Coronary Syndrome (NSTE-ACS) Patients
Acronym: ILLEPE-ACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Wei Feng Shen, Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJH-091228; RJH-2009 (Other: RuiJin Hospital, Shanghai Jiaotong University School of Medicine)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-02

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; intervention; outcome; patients diagnosed ad Non-ST elevation ACS; patients received PCI therapy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional group (Active Comparator): patients will be treated by atorvastation 20mg/d after randomization, and continued for one year.
  Interventions: Drug: Atorvastatin
- intensive group (Experimental): patient will be loaded with 80mg atorvastatin, continued by atorvastatin 40mg/d for 30d, then receive atorvastatin 20mg/d for the following 11 months.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — patients admitted for Non-ST elevation ACS will be treated by atorvastatin 20md/d for one year
  Arms: conventional group
Drug: Atorvastatin — patients admitted with Non-ST elevation ACS will be loaded with atorvastatin 80mg once, continued with 40mg/d for 30d, then change to 20mg/d, as a regular dose in China
  Arms: intensive group

SUMMARY:
PCI has been one of the most common choice of treatments for patients with coronary artery disease, and studies indicated that intensive statin treatment before PCI could reduce adverse events as comparing to the placebo. In China, statin with regular dose is currently applied to the patients admitted for Non-ST-elevation acute coronary syndrome (ACS). Here we hypothesize that intensive statin treatment with arovastatin before PCI could further reduce clinical adverse events.

ELIGIBILITY:
Inclusion Criteria:

* finish informed consent
* age≥18y and under 75y
* diagnosed as non-ST elevation acute coronary syndrome, including unstable angina and non-ST elevation myocardial infarction
* willing to receive the coronary angiography and potential PCI therapy

Exclusion Criteria:

* patient was treated by statins before randomization
* stable angina or ST elevation myocardial infarction
* without informed consent
* abnormal liver function before randomization, (AST，ALT≥3ULN)
* active hepatitis or muscular disease
* impaired renal function with serum creatinine level > 3mg/dl
* impaired left ventricular systolic function with LVEF< 30%
* participating in other studies
* non-PCI treated patients after coronary angiography will be washed out

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
The primary end point was the composite of major adverse cardiac events (MACE), including cardiac death, non-fatal reinfarction, and target vessel revascularization (TVR) at one-year clinical follow-up after randomization. | one year

SECONDARY OUTCOMES:
rate of peri-procedural myocardial infarction | 30days
MACE at 30d after randomization 3. changes of left ventricular function at 30d after randomization | 30 days
changes of left ventricular function at 30d after randomization | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng Shen, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital, Dept. of Cardiology, Shanghai, Shanghai Municipality, China